CLINICAL TRIAL: NCT01932619
Title: The Influence of Storage Container and Defrost Process on Components in Breast Milk
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: C08178
Record Dates: First submitted 2013-08-21; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Human Milk

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples Without DNA — breast milk
Oversight: Data Monitoring Committee: No

SUMMARY:
Breast milk is best food for neonates and preterm infants. However many handling would be done if direct breastfeeding is not feasible, and it may result in nutrients change in human milk. We investigate the influence of storage in different containers and different thawing or heating methods on human milk nutrients.

ELIGIBILITY:
Inclusion Criteria:

* healthy mothers lactating during first year of their babies and have sufficient milk to donate

Exclusion Criteria:

* mothers who have insufficient milk for their babies
* mothers have major disease or on specific diet or drug which would affect breast milk composition

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy mothers lactating breast milk during first year of their babies
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
changes in nutrients of human milk after several processing | within first year of milk expression
  we measure the changes of nutrients, including fat, protein, lactose, energy, immunoglobulins, lactoferrin, leptin, and lysozyme in human milk after several processes, such as freezing, pasteurization, storage in different containers, thawing, and heat treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Neonatology, Department of Pediatrics, Taichung Veterans General Hospital, Taichung, Taiwan